CLINICAL TRIAL: NCT03971838
Title: Diabetes Prevention Programming for Women With a History of Gestational Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Tamara S. Hannon, Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 1812789354
Record Dates: First submitted 2019-05-24; First posted 2019-06-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Women with a history of gestational diabetes will be offered 4-6 months of a diabetes prevention program.
  Interventions: Behavioral: Positive Outcomes for Women

INTERVENTIONS:
Behavioral: Positive Outcomes for Women — Women and their children 10+ can consent to participate in the diabetes prevention programming offered through the research center. We will collect data at three time points, baseline, 4-6 months, and 12 months.
  2. Instead of participating in Encourage, women may participate in other diabetes prevention programming/weight management programming offered by other entities. Researchers will consent these women into the study to complete 3 data collection points, baseline, 4-6 months, and 12 months. Additionally, researchers will consent women to obtain data from their chosen program. For instance, if a woman chooses to do a Diabetes Prevention Program through the YMCA, researchers will ask women to self report their weekly attendance and weight.

SUMMARY:
The purpose of this study is to offer women with a history of gestational diabetes access to diabetes prevention programming; their children 10 and older can participate.

DETAILED DESCRIPTION:
The purpose of this study is to offer women with a history of gestational diabetes access to diabetes prevention programming; their children 10 and older can participate. There are two potential types of participants:

1. Women and their children 10+ can consent to participate in the diabetes prevention programming offered through Dr. Hannon's center (called Encourage). Researchers will collect data at three time points, baseline, 4-6 months, and 12 months.
2. Instead of participating in Encourage, women may participate in other diabetes prevention programming/weight management programming offered by other entities. Researchers will consent these women into the study to complete 3 data collection points, baseline, 4-6 months, and 12 months. Additionally, researchers will consent women to obtain data from their chosen program. For instance, if a woman chooses to do a Diabetes Prevention Program through the YMCA, researchers will ask women to self report their weekly attendance and weight.

ELIGIBILITY:
Inclusion Criteria:

* History of gestational diabetes in a previous pregnancy
* Age 18+

Exclusion Criteria:

·Currently pregnant

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 117 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Enrollment and participation rates in a diabetes prevention intervention | 12 months
  Enrollment and participation rates in a diabetes prevention intervention

SECONDARY OUTCOMES:
HbA1c | 12 months
  HbA1c
BMI | 12 months
  Height and weight combined to report as BMI

CONTACTS AND LOCATIONS:
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided
Undecided